CLINICAL TRIAL: NCT04150900
Title: 1922GCCC: PHASE 2 STUDY OF PEMBROLIZUMAB AND BAVITUXIMAB FOR PROGRESSIVE RECURRENT/METASTATIC SQUAMOUS CELL CARCINOMA OF THE HEAD AND NECK
Brief Title: 1922GCCC: Pembro and Bavituximab for Squamous Cell Carcinoma of Head and Neck
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1922GCCC_HP-00085668
Record Dates: First submitted 2019-10-22; First posted 2019-11-05 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-12

CONDITIONS: Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — bavituximab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Pembro and Bavituximab for progressive recurrent/metastatic squamous cell carcinoma of head and neck
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Bavituximab (Experimental): Pembro and Bavituximab for progressive recurrent/metastatic squamous cell carcinoma of head and neck
  Interventions: Drug: Bavituximab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Bavituximab — Bavituximab is a chimeric (human/mouse) monoclonal antibody (mAb) derived from murine mAb 3G4 that targets phosphatidylserine (PS) after binding to β2-glycoprotein 1 (β2-GP1).
Drug: Pembrolizumab — Pembrolizumab is a highly selective humanized mAb designed to block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.

SUMMARY:
This phase II single arm study is being done to determine if bavituximab could potentially synergize with PD-1 inhibitor therapy to generate an effective anti-tumor immune response in patients with recurrent/metastatic squamous cell head and neck cancer (HNSCC) who progressed on a PD-1 inhibitor.

DETAILED DESCRIPTION:
The goal of this study is to assess whether treatment with bavituximab shifts the cellular balance to favor an effective T-cell mediated antitumor response resulting to an enhanced response in conjunction with pembrolizumab. Bavituximab is a chimeric (human/mouse) monoclonal antibody that targets phosphatidylserine (PS). PS facilitates the recognition and clearance of dying cells, triggering the release of immunosuppressive cytokines and inhibiting the production of proinflammatory cytokines. Within the tumor microenvironment, PS polarizes macrophages toward an immunosuppressive phenotype. Bavituximab upregulates the adaptive T cell-mediated response through crosslinking FCRγ and dampening of signaling between PS and PS receptors on immunosuppressive myeloid-derived suppressor cells.

Thus, the investigators are doing this phase II single arm study to determine if bavituximab could potentially synergize with PD-1 inhibitor therapy to generate an effective anti-tumor immune response in patients with recurrent/metastatic squamous cell head and neck cancer (HNSCC) who progressed on a PD-1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have recurrent/metastatic head and neck cancer and will have radiographic evidence of progression on prior immune checkpoint inhibitor therapy, including nivolumab, pembrolizumab, durvalumab and atezolizumab. Patients must have progressed on prior platinum therapy either in the recurrent setting or within 6 months of treatment with cisplatin and radiation in the potentially curative setting.
* Be willing and able to provide written informed consent/assent for the trial.
* Be > or equal to 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the PI.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.
* Female subject of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential (Section 6.2) must be willing to use an adequate method of contraception as outlined in Section 6.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

-Male subjects of childbearing potential (Section 6.2) must agree to use an adequate method of contraception as outlined in Section 6.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients. History of hypersensitivity to other antibodies can be discussed with the PI to determine eligibility.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

* Has experienced an immune-related adverse event requiring discontinuation of a prior checkpoint inhibitor.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement (such as prednisone 10mg daily or its equivalent) for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids and adrenal replacement steroid doses < 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.

Inclusion of Women and Minorities

Both men and women of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2027-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seiwert TY, Burtness B, Mehra R, Weiss J, Berger R, Eder JP, Heath K, McClanahan T, Lunceford J, Gause C, Cheng JD, Chow LQ. Safety and clinical activity of pembrolizumab for treatment of recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-012): an open-label, multicentre, phase 1b trial. Lancet Oncol. 2016 Jul;17(7):956-965. doi: 10.1016/S1470-2045(16)30066-3. Epub 2016 May 27. PMID 27247226
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Balermpas P, Rodel F, Rodel C, Krause M, Linge A, Lohaus F, Baumann M, Tinhofer I, Budach V, Gkika E, Stuschke M, Avlar M, Grosu AL, Abdollahi A, Debus J, Bayer C, Stangl S, Belka C, Pigorsch S, Multhoff G, Combs SE, Monnich D, Zips D, Fokas E. CD8+ tumour-infiltrating lymphocytes in relation to HPV status and clinical outcome in patients with head and neck cancer after postoperative chemoradiotherapy: A multicentre study of the German cancer consortium radiation oncology group (DKTK-ROG). Int J Cancer. 2016 Jan 1;138(1):171-81. doi: 10.1002/ijc.29683. Epub 2015 Jul 30. PMID 26178914
- [Background] Kim KJ, Lee KS, Cho HJ, Kim YH, Yang HK, Kim WH, Kang GH. Prognostic implications of tumor-infiltrating FoxP3+ regulatory T cells and CD8+ cytotoxic T cells in microsatellite-unstable gastric cancers. Hum Pathol. 2014 Feb;45(2):285-93. doi: 10.1016/j.humpath.2013.09.004. Epub 2013 Dec 12. PMID 24331841
- [Background] Savas P, Salgado R, Denkert C, Sotiriou C, Darcy PK, Smyth MJ, Loi S. Clinical relevance of host immunity in breast cancer: from TILs to the clinic. Nat Rev Clin Oncol. 2016 Apr;13(4):228-41. doi: 10.1038/nrclinonc.2015.215. Epub 2015 Dec 15. PMID 26667975
- [Background] Uppaluri R, Dunn GP, Lewis JS Jr. Focus on TILs: prognostic significance of tumor infiltrating lymphocytes in head and neck cancers. Cancer Immun. 2008 Dec 4;8:16. PMID 19053167
- [Background] Shinto E, Hase K, Hashiguchi Y, Sekizawa A, Ueno H, Shikina A, Kajiwara Y, Kobayashi H, Ishiguro M, Yamamoto J. CD8+ and FOXP3+ tumor-infiltrating T cells before and after chemoradiotherapy for rectal cancer. Ann Surg Oncol. 2014 Jun;21 Suppl 3:S414-21. doi: 10.1245/s10434-014-3584-y. Epub 2014 Feb 25. PMID 24566864
- [Background] Vassilakopoulou M, Avgeris M, Velcheti V, Kotoula V, Rampias T, Chatzopoulos K, Perisanidis C, Kontos CK, Giotakis AI, Scorilas A, Rimm D, Sasaki C, Fountzilas G, Psyrri A. Evaluation of PD-L1 Expression and Associated Tumor-Infiltrating Lymphocytes in Laryngeal Squamous Cell Carcinoma. Clin Cancer Res. 2016 Feb 1;22(3):704-13. doi: 10.1158/1078-0432.CCR-15-1543. Epub 2015 Sep 25. PMID 26408403
- [Background] Topalian SL, Taube JM, Anders RA, Pardoll DM. Mechanism-driven biomarkers to guide immune checkpoint blockade in cancer therapy. Nat Rev Cancer. 2016 May;16(5):275-87. doi: 10.1038/nrc.2016.36. Epub 2016 Apr 15. PMID 27079802
- [Background] Shinohara T, Taniwaki M, Ishida Y, Kawaichi M, Honjo T. Structure and chromosomal localization of the human PD-1 gene (PDCD1). Genomics. 1994 Oct;23(3):704-6. doi: 10.1006/geno.1994.1562. PMID 7851902
- [Background] Bertucci F, Finetti P, Mamessier E, Pantaleo MA, Astolfi A, Ostrowski J, Birnbaum D. PDL1 expression is an independent prognostic factor in localized GIST. Oncoimmunology. 2015 Feb 3;4(5):e1002729. doi: 10.1080/2162402X.2014.1002729. eCollection 2015 May. PMID 26155391
- [Background] Kim HR, Ha SJ, Hong MH, Heo SJ, Koh YW, Choi EC, Kim EK, Pyo KH, Jung I, Seo D, Choi J, Cho BC, Yoon SO. PD-L1 expression on immune cells, but not on tumor cells, is a favorable prognostic factor for head and neck cancer patients. Sci Rep. 2016 Nov 14;6:36956. doi: 10.1038/srep36956. PMID 27841362
- [Background] Mishra AK, Kadoishi T, Wang X, Driver E, Chen Z, Wang XJ, Wang JH. Squamous cell carcinomas escape immune surveillance via inducing chronic activation and exhaustion of CD8+ T Cells co-expressing PD-1 and LAG-3 inhibitory receptors. Oncotarget. 2016 Dec 6;7(49):81341-81356. doi: 10.18632/oncotarget.13228. PMID 27835902
- [Background] Mandal R, Senbabaoglu Y, Desrichard A, Havel JJ, Dalin MG, Riaz N, Lee KW, Ganly I, Hakimi AA, Chan TA, Morris LG. The head and neck cancer immune landscape and its immunotherapeutic implications. JCI Insight. 2016 Oct 20;1(17):e89829. doi: 10.1172/jci.insight.89829. PMID 27777979
- [Background] Balasubramanian K, Schroit AJ. Characterization of phosphatidylserine-dependent beta2-glycoprotein I macrophage interactions. Implications for apoptotic cell clearance by phagocytes. J Biol Chem. 1998 Oct 30;273(44):29272-7. doi: 10.1074/jbc.273.44.29272. PMID 9786940
- [Background] Soares MM, King SW, Thorpe PE. Targeting inside-out phosphatidylserine as a therapeutic strategy for viral diseases. Nat Med. 2008 Dec;14(12):1357-62. doi: 10.1038/nm.1885. Epub 2008 Nov 23. PMID 19029986
- [Background] Birge RB, Boeltz S, Kumar S, Carlson J, Wanderley J, Calianese D, Barcinski M, Brekken RA, Huang X, Hutchins JT, Freimark B, Empig C, Mercer J, Schroit AJ, Schett G, Herrmann M. Phosphatidylserine is a global immunosuppressive signal in efferocytosis, infectious disease, and cancer. Cell Death Differ. 2016 Jun;23(6):962-78. doi: 10.1038/cdd.2016.11. Epub 2016 Feb 26. PMID 26915293
- [Background] Yin Y, Huang X, Lynn KD, Thorpe PE. Phosphatidylserine-targeting antibody induces M1 macrophage polarization and promotes myeloid-derived suppressor cell differentiation. Cancer Immunol Res. 2013 Oct;1(4):256-68. doi: 10.1158/2326-6066.CIR-13-0073. Epub 2013 Aug 19. PMID 24777853
- [Background] Ran S, He J, Huang X, Soares M, Scothorn D, Thorpe PE. Antitumor effects of a monoclonal antibody that binds anionic phospholipids on the surface of tumor blood vessels in mice. Clin Cancer Res. 2005 Feb 15;11(4):1551-62. doi: 10.1158/1078-0432.CCR-04-1645. PMID 15746060
- [Background] DeRose P, Thorpe PE, Gerber DE. Development of bavituximab, a vascular targeting agent with immune-modulating properties, for lung cancer treatment. Immunotherapy. 2011 Aug;3(8):933-44. doi: 10.2217/imt.11.87. PMID 21843081
- [Background] Gerber DE, Hao G, Watkins L, Stafford JH, Anderson J, Holbein B, Oz OK, Mathews D, Thorpe PE, Hassan G, Kumar A, Brekken RA, Sun X. Tumor-specific targeting by Bavituximab, a phosphatidylserine-targeting monoclonal antibody with vascular targeting and immune modulating properties, in lung cancer xenografts. Am J Nucl Med Mol Imaging. 2015 Oct 12;5(5):493-503. eCollection 2015. PMID 26550540
- [Background] Bronte V, Serafini P, De Santo C, Marigo I, Tosello V, Mazzoni A, Segal DM, Staib C, Lowel M, Sutter G, Colombo MP, Zanovello P. IL-4-induced arginase 1 suppresses alloreactive T cells in tumor-bearing mice. J Immunol. 2003 Jan 1;170(1):270-8. doi: 10.4049/jimmunol.170.1.270. PMID 12496409
- [Background] Mazzoni A, Bronte V, Visintin A, Spitzer JH, Apolloni E, Serafini P, Zanovello P, Segal DM. Myeloid suppressor lines inhibit T cell responses by an NO-dependent mechanism. J Immunol. 2002 Jan 15;168(2):689-95. doi: 10.4049/jimmunol.168.2.689. PMID 11777962
- [Background] Corzo CA, Cotter MJ, Cheng P, Cheng F, Kusmartsev S, Sotomayor E, Padhya T, McCaffrey TV, McCaffrey JC, Gabrilovich DI. Mechanism regulating reactive oxygen species in tumor-induced myeloid-derived suppressor cells. J Immunol. 2009 May 1;182(9):5693-701. doi: 10.4049/jimmunol.0900092. PMID 19380816
- [Background] Identification of Myeloid-Dervied Suppressor cell sin squamous cell cancer of the head and neck. TrioMeetings.
- [Background] Horinaka A, Sakurai D, Ihara F, Makita Y, Kunii N, Motohashi S, Nakayama T, Okamoto Y. Invariant NKT cells are resistant to circulating CD15+ myeloid-derived suppressor cells in patients with head and neck cancer. Cancer Sci. 2016 Mar;107(3):207-16. doi: 10.1111/cas.12866. Epub 2016 Feb 13. PMID 26679292
- [Background] Freimark BD, Gong J, Ye D, Gray MJ, Nguyen V, Yin S, Hatch MM, Hughes CC, Schroit AJ, Hutchins JT, Brekken RA, Huang X. Antibody-Mediated Phosphatidylserine Blockade Enhances the Antitumor Responses to CTLA-4 and PD-1 Antibodies in Melanoma. Cancer Immunol Res. 2016 Jun;4(6):531-40. doi: 10.1158/2326-6066.CIR-15-0250. Epub 2016 Apr 4. PMID 27045021
- [Background] Huang X, Bennett M, Thorpe PE. A monoclonal antibody that binds anionic phospholipids on tumor blood vessels enhances the antitumor effect of docetaxel on human breast tumors in mice. Cancer Res. 2005 May 15;65(10):4408-16. doi: 10.1158/0008-5472.CAN-05-0031. PMID 15899833
- [Background] Beck AW, Luster TA, Miller AF, Holloway SE, Conner CR, Barnett CC, Thorpe PE, Fleming JB, Brekken RA. Combination of a monoclonal anti-phosphatidylserine antibody with gemcitabine strongly inhibits the growth and metastasis of orthotopic pancreatic tumors in mice. Int J Cancer. 2006 May 15;118(10):2639-43. doi: 10.1002/ijc.21684. PMID 16353142
- [Background] Gerber DE, Stopeck AT, Wong L, Rosen LS, Thorpe PE, Shan JS, Ibrahim NK. Phase I safety and pharmacokinetic study of bavituximab, a chimeric phosphatidylserine-targeting monoclonal antibody, in patients with advanced solid tumors. Clin Cancer Res. 2011 Nov 1;17(21):6888-96. doi: 10.1158/1078-0432.CCR-11-1074. Epub 2011 Oct 11. PMID 21989064
- [Background] Chalasani P, Marron M, Roe D, Clarke K, Iannone M, Livingston RB, Shan JS, Stopeck AT. A phase I clinical trial of bavituximab and paclitaxel in patients with HER2 negative metastatic breast cancer. Cancer Med. 2015 Jul;4(7):1051-9. doi: 10.1002/cam4.447. Epub 2015 Mar 31. PMID 25826750
- [Background] Tabagari D, Nemsadze G, Janjalia M, et al. Phase II study of bavituximab plus docetaxel in locally advanced or metastatic breast cancer. J Clin Oncol 2010; 28(15s) Abstract 1042.
- [Background] Yopp A, Singal A, Arriaga YE, et al. A phase II study of bavituximab and sorafenib in advanced hepatocellular carcinoma (HCC). 2015 Gastrointestinal Cancers Symposium; 2015.
- [Background] Patnaik A, Kang SP, Rasco D, Papadopoulos KP, Elassaiss-Schaap J, Beeram M, Drengler R, Chen C, Smith L, Espino G, Gergich K, Delgado L, Daud A, Lindia JA, Li XN, Pierce RH, Yearley JH, Wu D, Laterza O, Lehnert M, Iannone R, Tolcher AW. Phase I Study of Pembrolizumab (MK-3475; Anti-PD-1 Monoclonal Antibody) in Patients with Advanced Solid Tumors. Clin Cancer Res. 2015 Oct 1;21(19):4286-93. doi: 10.1158/1078-0432.CCR-14-2607. Epub 2015 May 14. PMID 25977344
- [Background] Chow LQM, Haddad R, Gupta S, Mahipal A, Mehra R, Tahara M, Berger R, Eder JP, Burtness B, Lee SH, Keam B, Kang H, Muro K, Weiss J, Geva R, Lin CC, Chung HC, Meister A, Dolled-Filhart M, Pathiraja K, Cheng JD, Seiwert TY. Antitumor Activity of Pembrolizumab in Biomarker-Unselected Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma: Results From the Phase Ib KEYNOTE-012 Expansion Cohort. J Clin Oncol. 2016 Nov 10;34(32):3838-3845. doi: 10.1200/JCO.2016.68.1478. Epub 2016 Sep 30. PMID 27646946
- [Result] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab + Bavituximab
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Bavituximab
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 67 [54 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: CR+PR
Description: overall response rate
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 55 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Bavituximab
Number analyzed (Participants) | 7
Participants
  Progressive Disease | 7
  Complete Response | 0

2. Secondary Outcome: Progression
Description: Progression free survival
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Bavituximab
Number analyzed (Participants) | 7
Participants
  Progressive Disease | 7
  Progression Free Survival | 0

3. Secondary Outcome: Disease Progression
Description: Number of participants with disease progression. For duration of response, CT imaging and RECIST criteria were reviewed to measure patient's response and time of that duration. One cycle is 21 days.
Time Frame: From date of randomization until the date of first documented progression up to 100 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Bavituximab
Number analyzed (Participants) | 7
Participants
  Progression prior to Cycle 2 | 1
  Progression at Cycle 2 | 2
  Progression at Cycle 3 | 3
  Progression at Cycle 4 | 1

4. Secondary Outcome: Survival
Description: Overall survival
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Bavituximab
Number analyzed (Participants) | 7
Participants
  Patient Expired | 6
  Outcome Unknown | 1

5. Secondary Outcome: Participants With Laboratory Correlates of Response
Description: Number of participants with laboratory correlates of response.
  The following outcomes are being measured:
  PD-L1 expression pre and post treatment Presence of TILs (tumor infiltrating lymphocytes) pre and post treatment Assessment of immune markers in pre-treatment fresh and post-treatment biopsies and blood.
  Assessment of genomics and tumor mutation burden in select patients.
  These outcome measures are determined through archival tumor tissue and next generation sequencing.
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Bavituximab
Number analyzed (Participants) | 7
Participants
  Laboratory correlates of response | 0
  No Laboratory correlates of response | 7

ADVERSE EVENTS:
Time Frame: 55 months
Arm/Group | Pembrolizumab + Bavituximab
All-Cause Mortality (participants affected / at risk) | 6/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Bavituximab (N=7)
Fatigue (General disorders) | 3
Back Pain (General disorders) | 1
Bilateral Lower limb edema (General disorders) | 1
Bleeding of lower lip (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Digital pain/rash (General disorders) | 1
Dizziness (General disorders) | 2
Dry Cough (General disorders) | 1
Dysegeusia (General disorders) | 1
Dysphagia (General disorders) | 1
Epistaxis (General disorders) | 1
Eye Irritation (General disorders) | 1
Facial Edema (General disorders) | 1
Fever (General disorders) | 1
Headache (General disorders) | 2
Hypergylcemia (Blood and lymphatic system disorders) | 1
Infection of lower lip (General disorders) | 1
Inflammation of lip (General disorders) | 1
Intermittent Fever (General disorders) | 1
Intermittent Non-Cardiac Chest pain (General disorders) | 1
Joint Pain (General disorders) | 1
Nausea (General disorders) | 2
Neuropathic Neck Pain (General disorders) | 1
non-Cardiac Upper chest wall pain (General disorders) | 1
Odynophagia (General disorders) | 1
Pharyngeal Cutaneous fistual (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Stomach Pain (General disorders) | 1
Weight loss (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT04150900/Prot_SAP_000.pdf